CLINICAL TRIAL: NCT06387940
Title: Investigation Into the Postprandial Effects of Varying Calorie Content of Low-Carbohydrate Diets on Human Metabolic Health
Brief Title: Acute Metabolic Effects of Carbohydrate Restriction at Varying Energy Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UEC 2019 008 FHMS
Record Dates: First submitted 2024-04-17; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal carbohydrate, energy-balanced diet, (nEB) (Active Comparator): provided participants' 100% daily energy needs, following the balanced Eatwell Guide recommendations.
  Interventions: Other: nEB Diet, followed for 36 hours
- low-carbohydrate, energy-balanced diet, (LCEB) (Active Comparator): diet contained just 50g of carbohydrates but still met 100% of the participants' estimated daily energy needs.
  Interventions: Other: LCEB Diet, followed for 36 hours
- low-carbohydrate, energy-restricted diet, (LC25) (Active Comparator): The diet consisted of only 50g of carbohydrates and provided 25% of the estimated daily energy needs.
  Interventions: Other: LC25 Diet, followed for 36 hours

INTERVENTIONS:
Other: nEB Diet, followed for 36 hours — nEB diet first, then LC25 and LCEB in random order with a 5 days washout between each diet
  Arms: normal carbohydrate, energy-balanced diet, (nEB)
Other: LC25 Diet, followed for 36 hours — LC25 diet first, then nEB and LCEB in random order with a 5 days washout between each diet
  Arms: low-carbohydrate, energy-restricted diet, (LC25)
Other: LCEB Diet, followed for 36 hours — LCEB diet first, then LC25 and nEB in random order with a 5 days washout between each diet
  Arms: low-carbohydrate, energy-balanced diet, (LCEB)

SUMMARY:
This study investigates how different low-carbohydrate diets affect metabolism and hunger in overweight adults. We will measure metabolic rates and blood metabolites.

DETAILED DESCRIPTION:
Participants will engage in three distinct eating plans: a standard diet with usual carbohydrate and calorie levels, a low-carb diet with typical calories, and a low-carb diet with reduced calories. Each diet is followed for a single day, with subsequent monitoring to assess how the body processes food and manages hunger after a meal. The goal is to understand the potential metabolic benefits of reducing carbohydrate intake, either alone or in combination with calorie reduction. This research aims to identify simpler dietary strategies that could improve heart health and assist in weight management without the need for severe calorie restriction or fasting, offering valuable insights for enhancing health outcomes in overweight individuals.

ELIGIBILITY:
Inclusion Criteria:

* stable weight within ±3 kg over the past three months
* no significant medical history.

Exclusion Criteria:

* pregnancy
* breastfeeding,
* using medications that could affect the study's outcomes
* high intake of caffeine and alcohol
* existing eating or psychiatric disorders
* adherence to strict dietary regimens like veganism
* high BMI resulting from significant muscle mass

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Biomarkers in blood Measured | 8 hours (fasting and post-meal)
  Measured with ELISA assay and clinical analyser (INDIKO)
Resting metabolic rate | 8 hours (fasting and post-meal)
  Measured with indirect calorimetry (GEM)

SECONDARY OUTCOMES:
Perceived Appetite Scores | 8 hours (fasting and post-meal)
  Measured with a Visual Analog Scale
Food intake | baseline and after each diet arm for 1 day
  Measured using food diaries

CONTACTS AND LOCATIONS:
Overall Officials: Hayriye Biyikoglu, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No